CLINICAL TRIAL: NCT01661049
Title: 1997-2011 Duodenal Cancer Analysis in Southern Denmark
Brief Title: Duodenal Cancer - Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Buchbjerg, Doctor, Odense University Hospital
Other Study IDs: 090377
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Duodenal Cancer
MeSH Terms: conditions — Duodenal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To see how a cohorte of 55 patients over periode 1997-2011 were mannaged, treated and survived duodenal cancer. Also to see how advanced the tumors were at time of diagnose and at time of operation.

ELIGIBILITY:
Inclusion Criteria:

* duodenal cancer

Exclusion Criteria:

* other cancers of the upper GI tract such as pancreatic cancer,
* cholangiocarcinoma,
* papilla Vateri cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with duodenal cancer
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2012-03

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Buchbjerg, Odense, Denmark